CLINICAL TRIAL: NCT05331742
Title: Comparison of Clinical Outcome Among Vaccinated and Unvaccinated Coronavirus Disease Patients Admitted to Critical Care Unit in a Tertiary Care Hospital of Kathmandu, Nepal.
Brief Title: Comparison of Clinical Outcome Among Vaccinated and Unvaccinated Coronavirus Disease Patients in Critical Care Unit.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Civil Service Hospital of Nepal (Other Government)
Responsible Party: Principal Investigator, Dr Deepak Bhandari, Registrar, Civil Service Hospital of Nepal
Other Study IDs: CSHNepal
Record Dates: First submitted 2022-04-08; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Coronavirus Infections; Critical Illness
MeSH Terms: conditions — Coronavirus Infections; Critical Illness | interventions — Vaccines

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vaccinated: patient between age 18 and above who have received a complete dose of coronavirus disease vaccine patient who has been admitted to critical care unit due to corona virus disease infection
  Interventions: Drug: Vaccine
- unvaccinated: patients between age 18 and above who has been admitted to critical care unit due to coronavirus disease infection and admitted to critical care unit

INTERVENTIONS:
Drug: Vaccine — patients who have received vaccine against coronavirus disease infection
  Groups: vaccinated

SUMMARY:
Corona virus disease has been a pandemic since its beginning. The problem has scaled to break health care system of multiple countries. One of the prime strategy of preventing this disease has been large mass scale vaccination campaign ongoing worldwide. No vaccine has been proven to 100 percent effective in preventing the infection with coronavirus disease so far. The investigators are conducting a study comparing outcome among vaccinated and unvaccinated population admitted to critical care unit of civil services hospital, Kathmandu , Nepal .

DETAILED DESCRIPTION:
Coronavirus disease has been a pandemic since its beginning. The problem has scaled up and health care system of multiple countries have reached to a breaking point . One of the prime strategy of preventing this disease has been large mass scale vaccination campaign ongoing worldwide. No vaccine has been proven to 100 percent effective in preventing the infection with coronavirus disease so far. The investigators are conducting a study comparing difference in outcome with regard to mortality and length of critical care unit stay among vaccinated and unvaccinated population admitted to critical care unit of civil services hospital , Kathmandu , Nepal.

Since different groups of population received different vaccine according to age profession and other factors investigators are trying to study the effectiveness of vaccine with regards to type of vaccine.

ELIGIBILITY:
Inclusion Criteria:

patients proven to have covid 19 infection patients more than 18 years of age patients admitted to critical care unit

Exclusion Criteria:

* patient below 18 years of age patients who do not have covid 19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients who had covid 19 infection and have been admitted to critical care unit will be enrolled in the study.
  Patient who have received vaccination against covid 19 infection yet are covid positive will be compared with patients who have not received covid 19 infection and have active covid 19 infection
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | within 12 weeks from the date of critical care unit admission
  the primary outcome to be measured will be difference in mortality among two groups (vaccinated and unvaccinated) of coronavirus infected patients admitted in critical care unit
length of icu stay | with 12 weeks from the date of critical care unit admission
  difference in length of stay between vaccinated and unvaccinated population admitted to critical care unit after being infected with coronavirus disease

SECONDARY OUTCOMES:
difference in mortality due to associated co-morbidity | within 24 weeks form the date of critical care unit admission
  difference in mortality due to associated co-morbidity will be compared among both the group (vaccinated and unvaccinated)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Bhandari, MD, Principal Investigator — Civil Services hospital , Kathmandu Nepal